CLINICAL TRIAL: NCT00539292
Title: A Multi-Centre, Prospective Randomized Trial to Evaluate Routine Use of a Silastic Spring-Loaded Silo for Infants With Gastroschisis
Brief Title: Evaluating the Use of a Silastic Spring-Loaded Silo for Infants With Gastroschisis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: With the existing rate of patient accrual, it would take an extensive amount of time to reach the initial target of 88 patients. During this period, other changes in perioperative management of surgical neonates may invalidate the study comparisons.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jacob Langer, Staff Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0020010078
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Gastroschisis
Keywords: pediatrics; gastroschisis; silastic spring-loaded silo
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Silastic Spring-Loaded Silo
  Interventions: Procedure: Primary placement of a spring-loaded silo
- 2 (Active Comparator): Primary Closure of Abdomen
  Interventions: Procedure: Primary Closure

INTERVENTIONS:
Procedure: Primary placement of a spring-loaded silo
  Arms: 1
Procedure: Primary Closure — primary closure of abdomen
  Arms: 2

SUMMARY:
This study seeks to evaluate whether the routine, primary use of the spring-loaded silo (SLS) to treat infants with gastroschisis will result in improved outcomes, faster recovery times and fewer post-surgical complications than the standard selective use of the silo.

DETAILED DESCRIPTION:
Standard treatment of the infant with gastroschisis consists of , the bowel being reduced into the abdomen, when possible,and the abdominal wall defect being closed in the operating room. When complete reduction of the eviscerated contents is not possible, a silastic " silo" is sewn on the abdominal wall and its contents are gradually reduced into the abdomen over several days. Once reduction is obtained, the silo is removed and the abdominal defect is closed.

Current methods of treatment are associated with significant morbidity, prolonged hospitalization, and high costs. Gastroschisis closure continues to be accompanied by a number of complications ranging from ileus, sepsis, TPN-related liver damage, necrotizing enterocolitis, respiratory insufficiency, and death. The optimal timing and method of closure, including primary versus secondary closure, continues to be debated. No prospective randomized studies to date have examined the routine use of the spring-loaded silo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gastroschisis
* Birth Weight ≥ 1500 grams
* Gestational Age ≥ 34 weeks

Exclusion Criteria:

* Birth Weight < 1500 grams
* Gestational Age < 34 weeks
* Presence of Bowel Ischemia or Necrosis
* Abdominal wall defect too small
* Major associated anomalies or medical condition
* Presence of Intracranial Hemorrhage (grade IV)
* Parent Refusal for Randomization

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Langer, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Pastor AC, Phillips JD, Fenton SJ, Meyers RL, Lamm AW, Raval MV, Lehman E, Karp TB, Wales PW, Langer JC. Routine use of a SILASTIC spring-loaded silo for infants with gastroschisis: a multicenter randomized controlled trial. J Pediatr Surg. 2008 Oct;43(10):1807-12. doi: 10.1016/j.jpedsurg.2008.04.003. PMID 18926212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 195 infants with gastroschisis were admitted to the participating centers between June 2001 and December 2006. After screening for eligibility and obtaining consent for enrollment, 55 patients were randomized. A randomization plan was generated by the lead center through an electronic Web-based randomization program.
Pre-assignment Details: 55 patients were randomized, 28 infants in the spring-loaded silo group and 27 infants in the primary closure group. One patient in the spring-loaded silo group was excluded from the study because of repeated dislodg-ement of the silo, requiring use of a sewn prosthetic device and inability to perform secondary closure.
Groups:
- Silastic Spring-Loaded Silo Group: Silastic Spring-Loaded Silo Group - Primary placement of a spring-loaded silo: routine bedside placement of a preformed Silastic spring-loaded silo, with gradual reduction and elective abdominal wall closure.
  Patients were assigned to 1 of the 2 groups using the sealed-envelope method.
  28 Infants had a spring-loaded silo placed in the delivery room or the neonatal intensive care unit. Reduction of the eviscerated bowel was accomplished by the daily application of gentle pressure, followed by the placement of a clip or umbilical tape across the silo to maintain the reduction. When the bowel was completely reduced, a clinical decision was made by the responsible surgeon for either silo removal and abdominal wall closure in the operating room under general anesthesia or abdominal wall closure at the bedside using the umbilical flap technique.
- Primary Closure of Abdomen Group: Primary Closure of Abdomen Group - Primary Closure: primary closure of abdomen: immediate attempt at primary closure, with placement of a silo only if primary closure was unsuccessful.
  Patients were assigned to 1 of the 2 groups using the sealed-envelope method.
  27 Infants underwent an attempt at primary closure. These infants underwent complete bowel reduction and abdominal wall closure, either in the operating room under general anesthesia or at the bedside. If the operating surgeon believed that primary closure would result in excessive lAP, a clinical decision was made to delay abdominal wall closure, and a spring-loaded silo was applied for gradual reduction and subsequent closure.
Period: Overall Study
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Started | 28 | 27
Completed | 27 | 27
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated in December 2006 (despite not achieving the initial target of 88 patients), the existing rate of patient accrual, would take an extensive amount of time to enter a planned number of patients; and during this period, other changes in perioperative management of surgical neonates may invalidate the study comparisons.
Groups:
- Silastic Spring-Loaded Silo Group: Silastic Spring-Loaded Silo Group
  Primary placement of a spring-loaded silo
  Silastic Spring-Loaded Silo Group - Primary placement of a spring-loaded silo: routine bedside placement of a preformed Silastic spring-loaded silo, with gradual reduction and elective abdominal wall closure.
  Patients were assigned to 1 of the 2 groups using the sealed-envelope method. 28 Infants had a spring-loaded silo placed in the delivery room or the neonatal intensive care unit. Reduction of the eviscerated bowel was accomplished by the daily application of gentle pressure, followed by the placement of a clip or umbilical tape across the silo to maintain the reduction. When the bowel was completely reduced, a clinical decision was made by the responsible surgeon for either silo removal and abdominal wall closure in the operating room under general anesthesia or abdominal wall closure at the bedside using the umbilical flap technique.
- Primary Closure of Abdomen Group: Primary Closure of Abdomen Group
  Primary Closure: primary closure of abdomen
  Primary Closure of Abdomen Group - Primary Closure: primary closure of abdomen: immediate attempt at primary closure, with placement of a silo only if primary closure was unsuccessful.
  Patients were assigned to 1 of the 2 groups using the sealed-envelope method. 27 Infants underwent an attempt at primary closure. These infants underwent complete bowel reduction and abdominal wall closure, either in the operating room under general anesthesia or at the bedside. If the operating surgeon believed that primary closure would result in excessive lAP, a clinical decision was made to delay abdominal wall closure, and a spring-loaded silo was applied for gradual reduction and subsequent closure.
- Total: Total of all reporting groups
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age (wk)
  weeks | 36.4 (1.2) | 36.7 (1.0) | 36.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 9 | 15 | 24
Birth weight (g) [Mean (Standard Deviation); unit: grams] | 2446 (567) | 2382 (391) | 2414 (479)

OUTCOME MEASURES:

1. Primary Outcome: Ventilation Status
Description: length of time on the ventilator
Time Frame: Data collected daily during the first 14 days after the abdominal wall closure (measured in days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Number analyzed (Participants) | 27 | 27
days | 3.17 (2.9) | 5.29 (5.2)

2. Secondary Outcome: Intraabdominal Pressure (IAP) as Reflected by Intragastric Pressure
Time Frame: intraabdominal pressure at the time of definitive closure
Population: The analysis of lAP at the time of abdominal wall closure was subject to adjustment as the data measured by intragastric catheter were only available for 15 patients in the spring-loaded silo group and 19 patients in the primary closure group.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Number analyzed (Participants) | 15 | 19
mm Hg | 10.9 (7) | 14.7 (5)

3. Secondary Outcome: TPN
Description: use of total parenteral nutrition (TPN)
Time Frame: Data collected daily during the first 14 days after the abdominal wall closure, then monthly for 3 months until discharge (measured in days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Number analyzed (Participants) | 27 | 27
days | 38.8 (33) | 33 (27)

4. Secondary Outcome: Length of Hospital Stay
Description: days in hospital
Time Frame: Data collected daily during the first 14 days after the abdominal wall closure (measured in days), then monthly for 3 months until discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Number analyzed (Participants) | 27 | 27
days | 49.1 (34) | 43.2 (28)

5. Secondary Outcome: Complications During Hospitalization (e.g., Sepsis)
Description: Clinical sepsis confirmed with a positive blood culture
Time Frame: post-surgery to hospital discharge; Data collected daily during the first 14 days after the abdominal wall closure (measured in days), then monthly for 3 months until discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
Number analyzed (Participants) | 27 | 27
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: Data collected daily during the first 14 days after the abdominal wall closure, then monthly for 3 months until discharge (measured in days)
Arm/Group | Silastic Spring-Loaded Silo Group | Primary Closure of Abdomen Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/27
Other Adverse Events (participants affected / at risk) | 2/27 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silastic Spring-Loaded Silo Group (N=27) | Primary Closure of Abdomen Group (N=27)
Short Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silastic Spring-Loaded Silo Group (N=27) | Primary Closure of Abdomen Group (N=27)
Atresia (Gastrointestinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Difficulty with patient enrollment because of parent refusal or absence for consent and individual surgeon preference not to randomize patients; this limited the number of patients enrolled and prevented adequate statistical power to be achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No